CLINICAL TRIAL: NCT04942132
Title: Managing Chronic Widespread Pain With FIBROLINE
Brief Title: Chronic Widespread Pain
Acronym: FIBROLINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Rovira i Virgili (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Obra Social de La Caixa (Unknown)
Responsible Party: Principal Investigator, Jordi Miró, Professor, University Rovira i Virgili
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSI2012-32471
Record Dates: First submitted 2017-01-11; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Mobile Health; Adolescents; Young adults; Fibromyalgia; Chronic Widespread Pain
MeSH Terms: conditions — Chronic Pain; Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): A Smartphone self-administered cognitive-behavioral based intervention
  Interventions: Behavioral: Cognitive-behavioral (CBT)

INTERVENTIONS:
Behavioral: Cognitive-behavioral (CBT) — Treatment includes a smartphone-delivered CBT program designed to improve the quality of life of individuals with chronic pain. The treatment is condensed in nine weeks, and contains the following modules or units of treatment: sleep quality, anxiety management, pain coping, medication use, physical conditioning, mood regulation, problem solving, decision-making and relationships with others. All the content and settings are written in Spanish.

SUMMARY:
Cognitive-behavioral treatments have proven effective in helping people with chronic pain. However, due to the limited availability of trained clinicians, many young people with chronic pain problems do not benefit from them. In order to overcome the shortage of clinicians researchers have begun to develop treatment programs that could be self-administered by smartphones. Although this is a step in the right direction, it is equally true that it also encloses a problematic issue. Namely, a large number of experienced clinicians would still be needed to oversee the functioning of these programs, and it does not seem likely that they will be available within a short time, at least in certain countries.

The objectives of this project are (1) to develop a web platform (iPAINs) to assist the clinician in the process of (a) creating and (b) administering cognitive-behavioral treatments for the management of chronic pain in adolescents and young adults, and (2) study the efficacy of a self-administered cognitive-behavioral treatment for young people with fibromyalgia or chronic widespread pain, developed and administered through iPAINs.

DETAILED DESCRIPTION:
iPAINs, will be a computer assisted device made to help create cognitive-behavioral treatment programs (and manage them) that can assist novice or expert professionals in the management of chronic pain in youths (experts who otherwise would not have the resources to develop and manage treatments via Smartphones). Therefore, it will help in the process of knowledge translation in this understudied and undertreated problem (of chronic pain in youths).

This platform (which includes an editor and administrator of treatments) will be evaluated in a sequential phased approach, consisting of 5 independent studies: (1) development of the tool and its contents (ie, digital objects of treatment), and (2) the web environment that allows creating and editing clinical treatments, (3) usability testing of iPAINs by a group of novice clinicians, and (4) experts clinicians to refine the prototype, and (5) a pilot study to determine the feasibility and effectiveness of the tool, that is, implementing a cognitive-behavioral self-administered treatment -through iPAINs- with patients with fibromyalgia or chronic widespread pain (Fibroline).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia or chronic widespread pain
* Capable of understanding, reading and writing in Spanish

Exclusion Criteria:

* Physical disabilities that interfered in the use of a Smartphone
* Severe cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Average Pain Intensity | through study completion, an average of 1 year
  Participants are asked to report three domains of pain intensity (i.e., average, worst, and current) using 0-10 numerical rating scales (NRS-11) with 0 meaning "No pain" and 10 meaning "Very much pain". A composite score (consisting of the mean of the individuals' three pain intensity scores) will be used as a measure of pain intensity.
Sleep Quality | through study completion, an average of 1 year
  Questionnaire used: Pittsburgh Sleep Quality Index (PSQI). The PSQI assesses sleep quality over the past month. The responder is requested to answer 19 questions that assess a variety of factors related to sleep quality. These 19 items generate seven component scores (each weighted equally on a 0-3 scale): sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medication and daytime dysfunction. The seven component scores are summed into a global PSQI score, which has a range of 0-21; higher score indicates worse sleep quality. This questionnaire includes five questions for the roommate of the responder which are used for clinical information and will not be included in this study.
Anxiety | through study completion, an average of 1 year
  Questionnaire used: The Spanish version of Patient-Reported Outcomes Measurement the Information System short form for Anxiety (PROMIS Short Form v1.0 - Anxiety 8a).
  It has 8 items asking about the frequency of physiological arousal, somatic symptoms and concerns in the past week. Participants will be asked to rate the frequency with which they experienced 8 anxiety symptoms in the last 7 days using a 5-point Likert scale (1= "Never"; 2 = "Almost never"; 3 = "Sometimes"; 4 = "Often"; 5 = "Almost always"). PROMIS-Anxiety has shown to provide a reliable measure of anxiety symptoms with ethnically diverse groups
Depression | through study completion, an average of 1 year
  Questionnaire used: The Spanish version of the PROMIS short form for Depression (PROMIS Short Form v1.0 - Depression 8a). This scale consists of 8 items that assesses the frequency of affective and cognitive manifestations of depression in the past week. The PROMIS Short Form v1.0 has been shown to provide a reliable measure of depressive symptoms when used with women with fibromyalgia
Fatigue | through study completion, an average of 1 year
  Questionnaire used: the Silhouettes Fatigue Scale (SFS) The SFS is a visual scale that has six human silhouettes showing an increasing level of fatigue from left to right, from "no fatigue" to "a lot of fatigue". SFS has shown to provide valid and reliable information when used with adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Chair in Pediatric Pain - Universitat Rovira i Virgili, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Research group webpage — http://algos-dpsico.urv.cat/en/